CLINICAL TRIAL: NCT06820242
Title: Development and Feasibility of a Mind-Body Intervention to Improve Physical Activity for Patients With Chronic Hip Pain: Open Pilot (HIPS Study)
Brief Title: Open Pilot Trial of a Mind-Body Intervention for Patients With Chronic Hip Pain
Acronym: HIPS Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kate Jochimsen, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025P000305; 5K23AT011922-04 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hip Pain; Hip Pain Chronic; Mind-Body Therapies
Keywords: chronic hip pain; mind-body; mindfulness

STUDY DESIGN:
Intervention Model Description: NIH Stage Model for Behavioral Intervention Development
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIPS (Experimental): A 6-session mind-body intervention that teaches patients with chronic hip joint-related pain (HRP) coping skills (e.g., SMART goal-setting, coping thoughts, deep breathing, and progressive muscle relaxation) and pain education.
  Interventions: Behavioral: HIPS

INTERVENTIONS:
Behavioral: HIPS — HIPS is a 6-session (one 30-minute session per week) mind-body intervention delivered virtually via live video by a trained physical therapist (PT). Across these six 30-minute sessions, the HIPS intervention aims to teach relaxation and coping skills (e.g., SMART goal-setting, coping thoughts, deep breathing, and progressive muscle relaxation) and provides pain education.

SUMMARY:
The goal of this study is to conduct a feasibility open pilot study (N=5) of HIPS with virtual exit interviews among adult patients with chronic hip joint-related pain (HRP). We will use this mixed methods information to assess the feasibility, credibility, and acceptability of the HIPS intervention and optimize the program and study methodology in preparation for a pilot feasibility randomized control trial (RCT).

Deliverables: [1] Adapt and refine open pilot protocol, patient recruitment, provider training, and other study materials. [2] Assess the feasibility, acceptability, and credibility of HIPS in preparation for a future feasibility RCT.

DETAILED DESCRIPTION:
Aim: Conduct a feasibility open pilot study (N=5) of HIPS with virtual exit interviews among adult patients with chronic HRP. The ultimate goal of this research is to assess the feasibility, credibility, and acceptability of the HIPS intervention and optimize the program and study methodology in preparation for a pilot feasibility randomized control trial (RCT).

HIPS Intervention: HIPS is a 6-session (one 30-minute session per week) mind-body intervention delivered virtually via live-video by a trained physical therapist (PT). In addition to participating in the HIPS intervention, all participants will attend their prescribed physical therapy with a physical therapist of their choosing. To minimize variability in physical rehabilitation, we will send the physical therapist the Clinical Practice Guidelines, which outline a standard-of-care rehabilitation protocol. Across the six 30-minute sessions, the HIPS intervention aims to teach relaxation and coping skills (e.g., SMART goal-setting, coping thoughts, deep breathing, and progressive muscle relaxation) and provides pain education. After each session, the participant is instructed to set and meet a physical activity SMART goal for the coming week. Within the program manual will be a log where the participant may track their completion of home practice. Each week, participants will receive a survey to formally report their daily home practice data over the last 7 days.

Following program completion, there will be a one-time 30-minute virtual exit interview to elicit subject perceptions of HIPS and any recommendations to improve intervention quality. This information will be used to further adapt and optimize HIPS prior to future efficacy testing.

Assessments: Baseline (0 weeks), post-test (6 weeks), and 6-month follow-up (30 weeks) survey assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting with chronic (lasting ≥3 months) hip joint-related pain (HRP)
2. Age ≥18yr

   a. If ≥45yr, the physician will confirm no osteoarthritis via X-ray (Kellgren Lawrence [KL] grade 0-1)
3. Score ≥3 for current hip pain on the Pain Visual Analogue Scale (Pain VAS)
4. Exhibits poor psychosocial health by meeting ≥1 of the criteria listed below:

   1. Score ≥ 20 on the Pain Catastrophizing Scale (PCS)
   2. Score ≤ 40 on the Pain Self-Efficacy Questionnaire (PSEQ)
   3. Score ≥ 17 on the Tampa Scale for Kinesiophobia (TSK-11)
5. Exhibits sedentariness by meeting ≥1 of the criteria listed below:

   1. Physically active < 150mins/week according to the International Physical Activity Questionnaire (IPAQ)
   2. Hip pain interferes with ability to be physically active
   3. Dissatisfaction with current physical activity level

Exclusion Criteria:

1. Previous surgery on the symptomatic (painful) hip
2. Current pain referred from the lower back

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Scored Above the Midpoint on Each Subscale of the Credibility and Expectancy Questionnaire | Baseline (0 Weeks)
  Assessed using the Credibility and Expectancy Questionnaire which asks the participant to indicate how much they believe, right now, that the intervention they will receive will help manage their COP and related worry. Possible scores range from 3 to 27 for both the credibility and the expectancy subscales. Higher scores represent higher credibility and expectancy.
Proportion of Participants Who Scored Above the Midpoint on the Client Satisfaction Scale | Post-Test (6 Weeks)
  Measured using the Client Satisfaction Scale which assess participants' satisfaction with participation in the study. The score range is 0-12. Higher scores indicate greater satisfaction.
Feasibility of recruitment | Baseline (0 Weeks)
  The percent of eligible patients approached that agree to participate.
Rate at which program was accepted, measured by number of completed program sessions | Post-Test (6 Weeks)
  The proportion of participants who attend ≥4 of 6 sessions.
Feasibility of Assessments at Baseline | Baseline (0 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Feasibility of Assessments at Post-Test | Post-Test (6 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Feasibility of Assessments at Follow-Up | Follow-Up (30 Weeks)
  Rate of participant's completion of self-report measures, with no measures missing.
Adverse Events | Collected during intervention, an average of 6 weeks
  Any self-reported or observed negative events related to participation
Therapist adherence | Collected during intervention, an average of 6 weeks
  Rate of interventionist's delivering the programs by following the established session topics and practices
Proportion of participants who report symptom improvements as measured by the Global Rating of Change Scale | Post-Test (6 Weeks)
  The proportion of participants who report overall improvement on the Global Rating of Change Scale. This measure includes a single question asking the patient to rate their change with respect to their hip condition over the last 6 weeks. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (Pain-VAS) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A single-item scale measuring self-reported pain intensity. Scores on the Pain-VAS range from 0 (no pain) to 100 (worst pain imaginable) and higher scores equate to worse outcomes.
International Hip Outcome Tool (iHOT-12) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 12-item questionnaire to assess deficiencies with respect to outcome assessment for young, active patients with hip disorders. Total scores range from 0 to 100 and higher scores represent better quality of life
PROMIS Pain Interference - Short Form 6b | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 6-item measure assessing self-reported consequences of pain on relevant aspects of a person's life and including the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Scores range from 6 to 30 where higher scores equate to worse outcomes.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 32-item state-trait questionnaire to measure multiple dimensions of interception. Scores on item range from 0 to 5 and higher scores translate to better outcomes.
International Physical Activity Questionnaire (IPAQ) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 27-item self-reported measure assessing physical activity. Overall score on the IPAQ is calculated using responses to all questions. More physical activity translates to better outcomes.
Pain Catastrophizing Scale (PCS) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 13-item questionnaire assessing one's tendency to focus on pain-related thoughts and feel helpless and hopeless due to pain on a scale of 0 to 4. Total scores range from 0 to 25 and higher scores indicate higher pain catastrophizing (worse outcomes).
Tampa Kinesiophobia Scale (TSK) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  An 11-item questionnaire that assesses fear avoidance and fear of activity. Summary score of total responses with Minimum = 11 and Maximum = 44. Higher scores indicate higher kinesiophobia.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 10-item measure assessing the confidence people with ongoing pain have in performing activities while in pain. Each item is scored on a 7-point Likert scale where 0 (not at all confident) and 6 (completely confident). Total scores range from 0 to 60 and higher scores translate to better outcomes.
Whole Person Health Index (WPHI) | Baseline (0 Weeks), Post-Test (6 Weeks), Follow-Up (30 Weeks)
  A 9-item measure assessing self-reported overall well-being. Each item is rated on a 1-5-point scale (total scores ranging from 9 to 45), with higher scores indicating worse overall well-being.
Change in Step Count via the ActiGraph wGT3X-BTLE Accelerometer | Baseline (0 Weeks), Post-Test (6 Weeks)
  Measures the change in steps during the 7 days following the baseline assessment and 7 days preceding the post-test. Larger increase in activity translate to better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States